CLINICAL TRIAL: NCT04375514
Title: A Phase 1/2a Dose-Escalating Study to Evaluate the Safety, Tolerability and Pharmacokinetic Effects of ARO-ENaC in Normal Healthy Volunteers and Safety, Tolerability and Efficacy in Patients With Cystic Fibrosis
Brief Title: Study of ARO-ENaC in Healthy Volunteers and in Patients With Cystic Fibrosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROENaC1001
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis, Pulmonary
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (12):
- Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 (Experimental): Normal healthy volunteers receive double-blind ARO-ENaC 20 mg on Days 1, 2, 3
  Interventions: Drug: ARO-ENaC
- Normal Healthy Volunteer Cohort: Placebo for ARO-ENaC 20 mg, Days 1-3 (Placebo Comparator): Normal healthy volunteers receive double-blind placebo for ARO-ENaC 20 mg on Days 1, 2, 3
  Interventions: Drug: Placebo
- Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 (Experimental): Normal healthy volunteers receive double-blind ARO-ENaC 40 mg on Days 1, 2, 3
  Interventions: Drug: ARO-ENaC
- Normal Healthy Volunteer Cohort: Placebo for ARO-ENaC 40 mg, Days 1-3 (Placebo Comparator): Normal healthy volunteers receive double-blind placebo for ARO-ENaC 40 mg on Days 1, 2, 3
  Interventions: Drug: Placebo
- Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 (Experimental): Normal healthy volunteers receive double-blind ARO-ENaC 65 mg on Days 1, 2, 3
  Interventions: Drug: ARO-ENaC
- Normal Healthy Volunteer Cohort: Placebo for ARO-ENaC 65 mg, Days 1-3 (Placebo Comparator): Normal healthy volunteers receive double-blind placebo for ARO-ENaC 65 mg on Days 1, 2, 3
  Interventions: Drug: Placebo
- Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 (Experimental): Normal healthy volunteers receive double-blind ARO-ENaC 180 mg on Days 1, 2, 3
  Interventions: Drug: ARO-ENaC
- Normal Healthy Volunteer Cohort: Placebo for ARO-ENaC 180 mg, Days 1-3 (Placebo Comparator): Normal healthy volunteers receive double-blind placebo for ARO-ENaC 180 mg on Days 1, 2, 3
  Interventions: Drug: Placebo
- Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy (Experimental): Normal healthy volunteers receive double-blind ARO-ENaC 180 mg on Days 1, 2, 3 with the purpose of collecting bronchoscopic samples
  Interventions: Drug: ARO-ENaC
- Normal Healthy Volunteer Cohort: Placebo for ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy (Placebo Comparator): Normal healthy volunteers receive double-blind placebo for ARO-ENaC 180 mg on Days 1, 2, 3 to collect bronchoscopic samples
  Interventions: Drug: Placebo
- Cystic Fibrosis Cohort: ARO-ENaC 40 mg, Days 1-3, 22-24 (Experimental): Participants with cystic fibrosis receive double-blind ARO-ENaC 40 mg dosed on Days 1, 2, and 3, and 40 mg dosed on Days 22, 23, and 24
  Interventions: Drug: ARO-ENaC
- Cystic Fibrosis Cohort: Placebo (Placebo Comparator): Participants with cystic fibrosis receive double-blind placebo for ARO-ENaC 40 mg dosed on Days 1, 2, and 3, and Days 22, 23, and 24.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARO-ENaC — single or multiple doses of ARO-ENaC by inhalation of nebulized solution
  Arms: Cystic Fibrosis Cohort: ARO-ENaC 40 mg, Days 1-3, 22-24; Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3; Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy; Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3; Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3; Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3
Drug: Placebo — calculated volume of normal saline to match active treatment by inhalation of nebulized solution
  Arms: Cystic Fibrosis Cohort: Placebo; Normal Healthy Volunteer Cohort: Placebo for ARO-ENaC 180 mg, Days 1-3; Normal Healthy Volunteer Cohort: Placebo for ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy; Normal Healthy Volunteer Cohort: Placebo for ARO-ENaC 20 mg, Days 1-3; Normal Healthy Volunteer Cohort: Placebo for ARO-ENaC 40 mg, Days 1-3; Normal Healthy Volunteer Cohort: Placebo for ARO-ENaC 65 mg, Days 1-3

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics (PK) of single doses of ARO-ENaC in healthy adult volunteers; and to evaluate the safety, tolerability, PK and efficacy of multiple doses of ARO-ENaC in patients with pulmonary cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be willing to use contraception
* Willing to provide written informed consent and to comply with study requirements
* Normal electrocardiogram (ECG) at Screening
* Non-smoking
* Normal pulmonary function tests at Screening (NHVs only)
* No abnormal finding of clinical relevance at Screening other than CF for CF patients
* Confirmed diagnosis of CF based on source verifiable medical record (CF patients only)
* All other treatments for CF have been stable for at least 2 months and patient is willing to continue this treatment regimen without change for duration of study (CF patients only)

Exclusion Criteria:

* Acute lower respiratory infection within 30 days of Screening (NHVs only)
* History of asthma (specifically, those subjects at risk of bronchial hyperactivity), anaphylaxis or airway hyper-reactivity
* Clinically significant history of hyperkalemia or presence of hyperkalemia at Screening
* Clinically significant health concerns (other than CF in CF patients)
* Human Immunodeficiency virus (HIV) infection, seropositive for Hepatitis B Virus (HBV), seropositive for Hepatitis C Virus (HCV)
* Uncontrolled hypertension
* Excessive use of alcohol within one month prior to Screening
* Use of illicit drugs within 1 year prior to Screening
* Use of an investigational agent or device within 30 days prior to dosing or current participation in an investigational study
* CF exacerbation within 30 days of Dosing (CF patients)
* History of solid organ transplant (CF patients)
* Diagnosis of hepatic cirrhosis (CF patients)

Note: additional inclusion/exclusion criteria may apply per protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2022-05-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (4):
  - Research Site 3, Chermside, Queensland
  - Research Site 4, South Brisbane, Queensland
  - Research Site 1, Nedlands, Washington
  - Research Site 2, Hamilton
- New Zealand (3):
  - Research Site 6, Grafton, Auckland
  - Research Site 8, Christchurch
  - Research Site 7, Dunedin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following Screening, eligible normal healthy volunteer participants enrolled and were randomly assigned 2:1 to receive ARO-ENaC or placebo on Days 1-3. Per protocol, the placebo cohorts were pooled for data analysis. Participants with cystic fibrosis were randomly assigned 2:1 to receive ARO-ENaC or placebo dosed on Days 1, 2, and 3, and Days 22, 23, and 24.
Groups:
- Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3: Normal healthy volunteers received double-blind ARO-ENaC 20 mg on Days 1, 2, 3
- Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3: Normal healthy volunteers received double-blind ARO-ENaC 40 mg on Days 1, 2, 3
- Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3: Normal healthy volunteers received double-blind ARO-ENaC 65 mg on Days 1, 2, 3
- Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3: Normal healthy volunteers received double-blind ARO-ENaC 180 mg on Days 1, 2, 3
- Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy: Normal healthy volunteers receive double-blind ARO-ENaC 180 mg on Days 1, 2, 3 to collect bronchoscopic samples before and after dosing.
- Normal Healthy Volunteer Cohort: Pooled Placebo: Normal healthy volunteers received double-blind sterile normal saline (0.9% NaCl) on Days 1, 2, 3
- Cystic Fibrosis Cohort: ARO-ENaC 40 mg, Days 1-3, 22-24: Participants with cystic fibrosis received double-blind ARO-ENaC 40 mg dosed on Days 1, 2, and 3, and 40 mg dosed on Days 22, 23, and 24.
- Cystic Fibrosis Cohort: Placebo: Participants with cystic fibrosis received double-blind placebo dosed on Days 1, 2, and 3, and Days 22, 23, and 24.
Period: Overall Study
Arm/Group | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy | Normal Healthy Volunteer Cohort: Pooled Placebo | Cystic Fibrosis Cohort: ARO-ENaC 40 mg, Days 1-3, 22-24 | Cystic Fibrosis Cohort: Placebo
Started | 4 | 4 | 4 | 4 | 8 | 12 | 4 | 3
Completed | 4 | 4 | 4 | 4 | 8 | 12 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy | Normal Healthy Volunteer Cohort: Pooled Placebo | Cystic Fibrosis Cohort: ARO-ENaC 40 mg, Days 1-3, 22-24 | Cystic Fibrosis Cohort: Placebo | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8 | 12 | 4 | 3 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 4 | 8 | 12 | 4 | 3 | 43
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3 | 2 | 2 | 8 | 2 | 3 | 23
  Male | 4 | 1 | 1 | 2 | 6 | 4 | 2 | 0 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  White | 2 | 2 | 3 | 2 | 5 | 7 | 4 | 3 | 28
  More than one race | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 3 | 3 | 2 | 2 | 3 | 7 | 4 | 3 | 27
  Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 3
  Other | 1 | 1 | 2 | 0 | 2 | 4 | 0 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Adverse event (AE)=any untoward medical occurrence that does not necessarily have to have a causal relationship with this treatment. Treatment-emergent AEs (TEAEs)=AEs with onset on or after administration of study drug through end of study. Serious adverse event (SAE)= an AE that results in death; is life-threatening; requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a medically important event or reaction.
Time Frame: Normal Healthy Volunteers: Up to 29 (+/- 2) days post-dose; Participants with cystic fibrosis (CF): Up to 113 (+/- 5) days post-dose
Population: Safety Set (all enrolled participants who received at least one dose of active drug or placebo)
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy | Normal Healthy Volunteer Cohort: Pooled Placebo | Cystic Fibrosis Cohort: ARO-ENaC 40 mg, Days 1-3, 22-24 | Cystic Fibrosis Cohort: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8 | 12 | 4 | 3
Participants
  Any AE | 3 | 2 | 3 | 3 | 6 | 10 | 3 | 3
  Any TEAE | 2 | 2 | 3 | 2 | 6 | 8 | 3 | 3
  Any Treatment-Related TEAE | 1 | 1 | 2 | 2 | 1 | 5 | 2 | 1
  Any SAE | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Any TE SAE | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Any Treatment-Related TE SAE | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Any AE Resulting in Study Drug Withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any AE Resulting in Study Discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any AE Resulting in Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Serum Electrolytes: Potassium, Sodium, Bicarbonate and Chloride
Time Frame: Normal Healthy Volunteers: Baseline, Days 2, 3, 4, 8, 15, 18, 29 ; Participants with CF: Baseline, Days 2, 3, 4, 15, 22, 23. 24, 29, 37, 57, 71, 85, 91, 113
Population: Safety Set: all enrolled participants who received at least one dose of active drug or placebo. Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy | Normal Healthy Volunteer Cohort: Pooled Placebo | Cystic Fibrosis Cohort: ARO-ENaC 40 mg, Days 1-3, 22-24 | Cystic Fibrosis Cohort: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8 | 12 | 4 | 3
mmol/L
  Potassium: Change at Day 2 | 0.18 (0.10) | 0.03 (0.15) | 0.20 (0.75) | 0.20 (0.14) | -0.10 (0.53) | 0.11 (0.24) | -0.05 (0.191) | -0.03 (0.153)
  Potassium: Change at Day 3 | -0.08 (0.29) | 0.15 (0.26) | -0.13 (0.43) | 0.13 (0.15) | 0.04 (0.57) | 0.14 (0.39) | -0.08 (0.330) | 0.13 (0.351)
  Potassium: Change at Day 4 | -0.20 (0.61) | 0.13 (0.10) | 0.03 (0.22) | 0.50 (0.54) | -0.11 (0.52) | 0.12 (0.32) | -0.03 (0.222) | 0.27 (0.513)
  Potassium: Change at Day 8: number analyzed (Participants) | 4 | 4 | 4 | 4 | 8 | 12 | 0 | 0
  Potassium: Change at Day 8 | -0.18 (0.56) | 0.43 (0.48) | -0.15 (0.38) | 0.28 (0.26) | -0.23 (0.31) | 0.03 (0.22) |  |
  Potassium: Change at Day 15: number analyzed (Participants) | 4 | 4 | 4 | 4 | 0 | 8 | 4 | 3
  Potassium: Change at Day 15 | 0.15 (0.49) | 0.18 (0.44) | -0.05 (0.52) | -0.08 (0.43) |  | -0.04 (0.15) | 0.10 (0.216) | -0.13 (0.231)
  Potassium: Change at Day 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 4 | 0 | 0
  Potassium: Change at Day 18 |  |  |  |  | -0.16 (0.50) | 0.20 (0.27) |  |
  Potassium: Change at Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Potassium: Change at Day 22 |  |  |  |  |  |  | -0.10 (0.245) | -0.27 (0.306)
  Potassium: Change at Day 23: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Potassium: Change at Day 23 |  |  |  |  |  |  | -0.05 (0.370) | -0.07 (0.153)
  Potassium: Change at Day 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Potassium: Change at Day 24 |  |  |  |  |  |  | -0.03 (0.171) | 0.07 (0.321)
  Potassium: Change at Day 29 | -0.15 (0.65) | 0.18 (0.45) | -0.33 (0.22) | 0.05 (0.17) | -0.09 (0.37) | 0.03 (0.24) | -0.05 (0.173) | 0.00 (0.300)
  Potassium: Change at Day 37: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Potassium: Change at Day 37 |  |  |  |  |  |  | 0.13 (0.330) | 0.07 (0.404)
  Potassium: Change at Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Potassium: Change at Day 57 |  |  |  |  |  |  | -0.05 (0.311) | -0.10 (0.200)
  Potassium: Change at Day 71: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Potassium: Change at Day 71 |  |  |  |  |  |  | 0.03 (0.275) | 0.10 (0.265)
  Potassium: Change at Day 85: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Potassium: Change at Day 85 |  |  |  |  |  |  | 0.10 (0.356) | -0.25 (0.071)
  Potassium: Change at Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
  Potassium: Change at Day 91 |  |  |  |  |  |  | 0.03 (0.403) | -0.10 (0.283)
  Potassium: Change at Day 113: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
  Potassium: Change at Day 113 |  |  |  |  |  |  | -0.03 (0.321) | 0.07 (0.153)
  Sodium: Change at Day 2 | 0.0 (1.4) | -0.8 (1.7) | 0.0 (1.4) | 1.5 (3.3) | 1.1 (1.5) | 0.3 (0.9) | -0.5 (1.91) | -1.3 (0.58)
  Sodium: Change at Day 3 | -0.3 (1.7) | 1.3 (1.7) | -1.0 (0.8) | -0.3 (2.9) | 0.9 (1.0) | -0.3 (1.6) | 1.0 (2.71) | 0.3 (4.04)
  Sodium: Change at Day 4 | -1.3 (1.5) | -0.3 (1.9) | 0.3 (2.2) | 5.0 (2.0) | 0.4 (1.4) | 0.8 (1.5) | 0.5 (1.73) | -0.7 (2.52)
  Sodium: Change at Day 8: number analyzed (Participants) | 4 | 4 | 4 | 4 | 8 | 12 | 0 | 0
  Sodium: Change at Day 8 | 2.0 (2.2) | 2.5 (1.7) | 0.5 (2.4) | 1.5 (1.3) | 2.0 (1.7) | -0.3 (1.9) |  |
  Sodium: Change at Day 15: number analyzed (Participants) | 4 | 4 | 4 | 4 | 0 | 8 | 4 | 3
  Sodium: Change at Day 15 | 0.8 (1.7) | 0.0 (2.6) | 0.0 (1.4) | -1.0 (3.3) |  | -0.6 (1.6) | -0.5 (0.58) | -1.3 (1.53)
  Sodium: Change at Day 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 4 | 0 | 0
  Sodium: Change at Day 18 |  |  |  |  | 2.5 (1.9) | 2.3 (2.4) |  |
  Sodium: Change at Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Sodium: Change at Day 22 |  |  |  |  |  |  | 1.0 (1.83) | 0.3 (3.21)
  Sodium: Change at Day 23: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Sodium: Change at Day 23 |  |  |  |  |  |  | 1.5 (2.38) | 0.7 (3.79)
  Sodium: Change at Day 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Sodium: Change at Day 24 |  |  |  |  |  |  | 2.0 (3.92) | 1.3 (5.77)
  Sodium: Change at Day 29 | -0.5 (1.7) | 1.8 (1.3) | -0.3 (1.3) | 1.5 (4.5) | 1.8 (2.6) | 0.6 (1.7) | -0.5 (1.91) | 0.0 (1.00)
  Sodium: Change at Day 37: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Sodium: Change at Day 37 |  |  |  |  |  |  | 0.0 (2.45) | -0.7 (1.53)
  Sodium: Change at Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Sodium: Change at Day 57 |  |  |  |  |  |  | 0.3 (2.22) | -1.3 (1.53)
  Sodium: Change at Day 71: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Sodium: Change at Day 71 |  |  |  |  |  |  | 1.3 (0.50) | -0.3 (0.58)
  Sodium: Change at Day 85: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
  Sodium: Change at Day 85 |  |  |  |  |  |  | 1.0 (1.15) | 0.0 (1.41)
  Sodium: Change at Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
  Sodium: Change at Day 91 |  |  |  |  |  |  | 1.0 (1.83) | 0.0 (1.41)
  Sodium: Change at Day 113: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
  Sodium: Change at Day 113 |  |  |  |  |  |  | -1.0 (2.65) | -2.0 (1.00)
  Bicarbonate: Change at Day 2 | 0.0 (0.8) | 0.0 (0.8) | 0.5 (1.7) | -4.8 (4.2) | 0.4 (1.8) | -0.3 (2.5) | 1.8 (1.71) | 0.7 (3.79)
  Bicarbonate: Change at Day 3 | -2.0 (0.8) | -0.5 (1.7) | 0.5 (1.0) | -1.0 (2.4) | 0.9 (1.4) | -0.3 (1.6) | -1.0 (2.16) | 0.7 (1.53)
  Bicarbonate: Change at Day 4 | -0.5 (0.6) | 1.3 (1.3) | 1.0 (0.8) | 0.0 (1.6) | 1.1 (1.4) | 0.2 (2.0) | 2.8 (2.50) | 1.3 (1.53)
  Bicarbonate: Change at Day 8: number analyzed (Participants) | 4 | 4 | 4 | 4 | 8 | 12 | 0 | 0
  Bicarbonate: Change at Day 8 | -0.8 (2.1) | 1.3 (1.0) | -0.3 (2.1) | 1.3 (1.3) | 1.9 (1.5) | 0.3 (1.9) |  |
  Bicarbonate: Change at Day 15: number analyzed (Participants) | 4 | 4 | 4 | 4 | 0 | 8 | 4 | 3
  Bicarbonate: Change at Day 15 | -0.3 (0.5) | 1.0 (1.2) | -0.3 (0.5) | -0.5 (1.3) |  | -1.0 (1.1) | 2.0 (1.41) | 0.7 (3.21)
  Bicarbonate: Change at Day 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 4 | 0 | 0
  Bicarbonate: Change at Day 18 |  |  |  |  | 1.3 (1.4) | 1.8 (1.5) |  |
  Bicarbonate: Change at Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Bicarbonate: Change at Day 22 |  |  |  |  |  |  | 1.3 (2.63) | 0.3 (1.53)
  Bicarbonate: Change at Day 23: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Bicarbonate: Change at Day 23 |  |  |  |  |  |  | 1.0 (1.41) | 0.7 (0.58)
  Bicarbonate: Change at Day 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Bicarbonate: Change at Day 24 |  |  |  |  |  |  | 1.3 (2.22) | -1.3 (5.13)
  Bicarbonate: Change at Day 29 | -0.5 (1.3) | 0.8 (1.0) | 0.0 (0.8) | -0.5 (1.0) | 1.1 (1.2) | 0.2 (1.9) | 1.8 (1.50) | 0.3 (1.53)
  Bicarbonate: Change at Day 37: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Bicarbonate: Change at Day 37 |  |  |  |  |  |  | 1.5 (2.65) | 0.0 (1.73)
  Bicarbonate: Change at Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Bicarbonate: Change at Day 57 |  |  |  |  |  |  | 2.0 (2.45) | 1.3 (3.21)
  Bicarbonate: Change at Day 71: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Bicarbonate: Change at Day 71 |  |  |  |  |  |  | 1.8 (1.71) | 1.7 (1.53)
  Bicarbonate: Change at Day 85: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
  Bicarbonate: Change at Day 85 |  |  |  |  |  |  | 2.0 (2.94) | 1.5 (3.54)
  Bicarbonate: Change at Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
  Bicarbonate: Change at Day 91 |  |  |  |  |  |  | 3.0 (2.83) | 2.5 (2.12)
  Bicarbonate: Change at Day 113: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
  Bicarbonate: Change at Day 113 |  |  |  |  |  |  | 2.3 (1.15) | 2.7 (2.08)
  Chloride: Change at Day 2 | 0.3 (1.0) | -1.0 (2.4) | 0.0 (0.8) | 1.0 (2.6) | -0.3 (1.3) | -0.2 (0.9) | -0.8 (1.26) | 1.0 (1.00)
  Chloride: Change at Day 3 | 0.3 (1.3) | 0.0 (1.8) | -1.3 (1.0) | 1.0 (2.9) | -0.1 (1.4) | -0.6 (1.2) | -0.5 (1.29) | -1.0 (2.00)
  Chloride: Change at Day 4 | -0.8 (0.5) | -2.8 (1.9) | -1.0 (1.4) | -0.5 (2.4) | -1.4 (1.8) | -0.6 (2.1) | 0.0 (1.41) | -2.0 (1.00)
  Chloride: Change at Day 8: number analyzed (Participants) | 4 | 4 | 4 | 4 | 8 | 12 | 0 | 0
  Chloride: Change at Day 8 | 3.3 (3.2) | 0.8 (1.9) | 0.5 (1.0) | 1.8 (1.5) | 0.1 (2.4) | 0.0 (1.8) |  |
  Chloride: Change at Day 15: number analyzed (Participants) | 4 | 4 | 4 | 4 | 0 | 8 | 4 | 3
  Chloride: Change at Day 15 | 2.3 (0.5) | -1.5 (2.6) | -0.3 (2.1) | 0.0 (3.3) |  | 0.6 (1.7) | -1.8 (2.22) | 0.7 (3.51)
  Chloride: Change at Day 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 12 | 0 | 0
  Chloride: Change at Day 18 |  |  |  |  | 1.0 (2.1) | -0.5 (1.7) |  |
  Chloride: Change at Day 22: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Chloride: Change at Day 22 |  |  |  |  |  |  | -1.3 (3.30) | 0.0 (1.00)
  Chloride: Change at Day 23: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Chloride: Change at Day 23 |  |  |  |  |  |  | -0.8 (3.50) | 1.3 (3.06)
  Chloride: Change at Day 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Chloride: Change at Day 24 |  |  |  |  |  |  | -0.5 (3.11) | 0.7 (5.03)
  Chloride: Change at Day 29 | 1.3 (1.9) | -0.5 (1.3) | 0.8 (0.5) | 0.8 (2.1) | -0.4 (2.6) | 0.6 (1.7) | -1.8 (3.30) | 0.7 (2.89)
  Chloride: Change at Day 37: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Chloride: Change at Day 37 |  |  |  |  |  |  | -2.0 (1.83) | 1.7 (4.04)
  Chloride: Change at Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Chloride: Change at Day 57 |  |  |  |  |  |  | -0.5 (2.38) | 1.3 (2.89)
  Chloride: Change at Day 71: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
  Chloride: Change at Day 71 |  |  |  |  |  |  | 0.8 (1.71) | 1.0 (1.73)
  Chloride: Change at Day 85: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
  Chloride: Change at Day 85 |  |  |  |  |  |  | 0.8 (1.71) | 1.5 (2.12)
  Chloride: Change at Day 91: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
  Chloride: Change at Day 91 |  |  |  |  |  |  | -1.0 (1.83) | 0.5 (0.71)
  Chloride: Change at Day 113: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
  Chloride: Change at Day 113 |  |  |  |  |  |  | 0.0 (3.00) | -1.7 (1.15)

3. Secondary Outcome: Change From Baseline in Forced Expiratory Volume (FEV1) in Normal Healthy Volunteers
Time Frame: Baseline, Up through Day 29 after a single dose
Population: Safety Set: all enrolled normal healthy volunteer participants who received at least one dose of active drug or placebo. Participants with an evaluable assessment at given time point.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy | Normal Healthy Volunteer Cohort: Pooled Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8 | 12
liters
  Change at Day 1: 15 mins post-dose | -0.128 (0.119) | 0.070 (0.184) | -0.015 (0.233) | -0.210 (0.175) | -0.194 (0.316) | -0.103 (0.151)
  Change at Day 1: 60 mins post-dose | -0.175 (0.180) | 0.175 (0.362) | 0.015 (0.139) | -0.088 (0.138) | -0.076 (0.197) | -0.074 (0.136)
  Change at Day 1: 120 mins post-dose | -0.033 (0.134) | 0.180 (0.286) | 0.180 (0.139) | -0.008 (0.017) | -0.055 (0.235) | -0.045 (0.165)
  Change at Day 2: Pre-dose | -0.033 (0.214) | 0.170 (0.311) | 0.138 (0.078) | -0.240 (0.189) | 0.055 (0.243) | -0.024 (0.130)
  Change at Day 2: 15 mins post-dose | -0.090 (0.130) | 0.158 (0.320) | 0.068 (0.100) | -0.285 (0.245) | -0.039 (0.290) | -0.107 (0.174)
  Change at Day 2: 60 mins post-dose | -0.118 (0.170) | 0.225 (0.303) | 0.138 (0.149) | -0.275 (0.290) | 0.003 (0.249) | -0.069 (0.125)
  Change at Day 2: 120 mins post-dose | -0.068 (0.194) | 0.165 (0.289) | 0.243 (0.131) | -0.275 (0.171) | 0.053 (0.428) | -0.015 (0.137)
  Change at Day 3: Pre-dose | 0.013 (0.098) | 0.210 (0.400) | 0.193 (0.134) | -0.158 (0.215) | 0.113 (0.352) | -0.049 (0.104)
  Change at Day 3: 15 mins post-dose | -0.090 (0.156) | 0.155 (0.324) | 0.130 (0.107) | -0.253 (0.317) | -0.028 (0.362) | -0.103 (0.139)
  Change at Day 3: 60 mins post-dose | -0.023 (0.159) | 0.190 (0.322) | 0.188 (0.164) | -0.078 (0.324) | 0.050 (0.370) | -0.068 (0.163)
  Change at Day 3: 120 mins post-dose | 0.010 (0.164) | 0.248 (0.333) | 0.260 (0.184) | -0.065 (0.179) | 0.088 (0.334) | -0.028 (0.167)
  Change at Day 4 | -0.093 (0.120) | 0.253 (0.376) | 0.293 (0.090) | -0.113 (0.185) | 0.158 (0.339) | -0.067 (0.191)
  Change at Day 8 | -0.090 (0.136) | 0.220 (0.411) | 0.160 (0.193) | 0.015 (0.232) | 0.070 (0.277) | -0.008 (0.190)
  Change at Day 15: number analyzed (Participants) | 4 | 4 | 4 | 4 | 0 | 8
  Change at Day 15 | -0.165 (0.299) | 0.190 (0.306) | 0.233 (0.079) | -0.133 (0.171) |  | -0.040 (0.131)
  Change at Day 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 4
  Change at Day 18 |  |  |  |  | 0.039 (0.323) | -0.408 (0.413)
  Change at Day 29/end of study (EOS)/end of treatment (ET) | -0.333 (0.252) | 0.183 (0.336) | 0.163 (0.112) | 0.000 (0.182) | 0.150 (0.241) | -0.027 (0.196)

4. Secondary Outcome: Pharmacokinetics (PK) of ARO-ENaC: Maximum Observed Plasma Concentration (Cmax) in Normal Healthy Volunteers
Time Frame: Day 1: Pre-dose, 30, 60, 120 mins and 4, 6, 8, 16 hours post-inhalation; Day 2: Pre-dose (Day 1, 24-hour timepoint), then 1, 2, 4 hours post-inhalation; Day 3: (Day 2, 24 hour timepoint), 30, 60, 120 mins, 4, 6, 8, 16, 24 (On Day 4), 48 (on Day 5)
Population: Normal healthy volunteers with ADS-003 plasma concentration above the lower limit of quantitation (LLOQ, 1.00 ng/mL). Participants who received placebo doses, all participants in ARO-ENaC 20 mg cohort, and 1 participant in the 40 mg cohort had plasma concentrations below the LLOQ. One participant in the 180 mg cohort had a single plasma sample, preventing the calculation of PK parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy | Normal Healthy Volunteer Cohort: Pooled Placebo
Number analyzed (Participants) | 0 | 3 | 4 | 3 | 8 | 0
ng/mL |  | 3.33 (1.6) | 8.37 (0.667) | 40.5 (16.1) | 56.7 (23.8) |

5. Secondary Outcome: PK of ARO-ENaC: Cmax in Participants With CF
Time Frame: Cycle 1 Day 1: Pre-dose (PrD), 30, 60, 120 minutes (m), 4 hours (h) post-dose (PoD); Day 2: PrD, 60, 120 m, 4 h PoD; Day 3: PrD, 30, 60, 120 m, 4 h PoD. Cycle 2 Days 22 and 23: PrD, 30 m, 4 h PoD; Day 24: PrD, 30, 60, 120 m, 4 h PoD
Population: Participants with CF with ADS-003 plasma concentration above the LLOQ (1.00 ng/mL). Participants who received placebo doses had plasma concentrations below the LLOQ. One participant had 3 plasma samples with concentrations close to the LLOQ preventing the calculation of PK parameters.
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Cystic Fibrosis Cohort: ARO-ENaC 40 mg, Days 1-3, 22-24 | Cystic Fibrosis Cohort: Placebo
Number analyzed (Participants) | 3 | 0
mg/mL
  Cycle 1 (Days 1 to 3) | 13.1 (8.9) |
  Cycle 2 (Days 22 to 24) | 9.8 (6.2) |

6. Secondary Outcome: PK of ARO-ENaC: Time to Maximum Plasma Concentration (Tmax) in Normal Healthy Volunteers
Time Frame: as for outcome 4
Population: Normal healthy volunteers with ADS-003 plasma concentration above the LLOQ (1.00 ng/mL). Participants who received placebo doses, all participants in ARO-ENaC 20 mg cohort, and 1 participant in the 40 mg cohort had plasma concentrations below the LLOQ. One participant in the 180 mg cohort had a single plasma sample, preventing the calculation of PK parameters.
Measure: Median (Full Range); unit: hours
Arm/Group | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy | Normal Healthy Volunteer Cohort: Pooled Placebo
Number analyzed (Participants) | 0 | 3 | 4 | 3 | 8 | 0
hours |  | 28 [4.0 to 52] | 39 [25 to 64] | 50 [50 to 54] | 2 [1 to 56] |

7. Secondary Outcome: PK of ARO-ENaC: Tmax in Participants With CF
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Cystic Fibrosis Cohort: ARO-ENaC 40 mg, Days 1-3, 22-24 | Cystic Fibrosis Cohort: Placebo
Number analyzed (Participants) | 3 | 0
hours
  Cycle 1 (Days 1 to 3) | 25 [0.5 to 49] |
  Cycle 2 (Day 22 to 24) | 25 [0.50 to 49.5] |

8. Secondary Outcome: PK of ARO-ENaC: Elimination Half-Life (t1/2) in Normal Healthy Volunteers
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy | Normal Healthy Volunteer Cohort: Pooled Placebo
Number analyzed (Participants) | 0 | 3 | 4 | 3 | 8 | 0
hours |  | 11 (1.2) | 10 (3.6) | 16 (3.0) | 10 (0.9) |

9. Secondary Outcome: PK of ARO-ENaC: Area Under the Plasma Concentration Versus Time Curve From Zero to the Last Quantifiable Plasma Concentration (AUClast) in Normal Healthy Volunteers
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h·mg/mL
Arm/Group | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy | Normal Healthy Volunteer Cohort: Pooled Placebo
Number analyzed (Participants) | 0 | 3 | 4 | 3 | 8 | 0
h·mg/mL |  | 91.7 (46.1) | 247 (106) | 1620 (577) | 1665 (650) |

10. Secondary Outcome: PK of ARO-ENaC: AUClast in Participants With CF
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h·mg/mL
Arm/Group | Cystic Fibrosis Cohort: ARO-ENaC 40 mg, Days 1-3, 22-24 | Cystic Fibrosis Cohort: Placebo
Number analyzed (Participants) | 3 | 0
h·mg/mL
  Cycle 1 (Days 1 to 3) | 155 (34.6) |
  Cycle 2 (Day 22 to 24) | 129 (47.7) |

11. Secondary Outcome: PK of ARO-ENaC: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUCinf) in Normal Healthy Volunteers
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h·mg/mL
Arm/Group | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy | Normal Healthy Volunteer Cohort: Pooled Placebo
Number analyzed (Participants) | 0 | 3 | 4 | 3 | 8 | 0
h·mg/mL |  | 117 (43.6) | 258 (145) | 1762 (668) | 1709 (660) |

12. Secondary Outcome: PK of ARO-ENaC: Plasma Clearance (CL/F) in Normal Healthy Volunteers
Time Frame: as for outcome 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy | Normal Healthy Volunteer Cohort: Pooled Placebo
Number analyzed (Participants) | 0 | 3 | 4 | 3 | 8 | 0
L/h |  | 227 (107) | 176 (85) | 75 (24) | 69 (20) |

13. Secondary Outcome: PK of ARO-ENaC: CL/F in Participants With CF
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cystic Fibrosis Cohort: ARO-ENaC 40 mg, Days 1-3, 22-24 | Cystic Fibrosis Cohort: Placebo
Number analyzed (Participants) | 3 | 0
L/h
  Cycle 1 (Days 1 to 3) | 101 (20) |
  Cycle 2 (Day 22 to 24) | 138 (46) |

14. Secondary Outcome: PK of ARO-ENaC: Amount Recovered in Urine Over 0 to 24 Hours Postdose (Ae0-24h) in Normal Healthy Volunteers
Time Frame: as for outcome 4
Population: Normal healthy volunteers in Cohorts 1-4 with ADS-003 plasma concentration above the LLOQ (1.00 ng/mL). Participants in ARO-ENaC 20 mg cohort, and 1 participant in the 40 mg cohort had plasma concentrations below the LLOQ. One participant in the 180 mg cohort had a single plasma sample, preventing the calculation of PK parameters.
Measure: Mean (Standard Deviation); unit: μg
Arm/Group | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3
Number analyzed (Participants) | 0 | 3 | 4 | 3
μg |  | 8.81 (2.55) | 22.0 (6.98) | 69.2 (8.30)

15. Secondary Outcome: PK of ARO-ENaC: Fraction Excreted in Urine as Unchanged Drug Over 0 to 24 Hours Postdose (fe0-24h) in Normal Healthy Volunteers
Time Frame: as for outcome 4
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: fraction of study drug
Arm/Group | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3
Number analyzed (Participants) | 0 | 3 | 4 | 3
fraction of study drug |  | 0.134 (0.0387) | 0.176 (0.0559) | 0.225 (0.0270)

16. Secondary Outcome: PK of ARO-ENaC: Renal Clearance (CLR) in Normal Healthy Volunteers
Time Frame: as for outcome 4
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3
Number analyzed (Participants) | 0 | 3 | 4 | 3
mL/h |  | 371 (262) | 210 (137) | 129 (54)

ADVERSE EVENTS:
Time Frame: Normal Healthy Volunteers: From Screening up to Day 29 ; CF Participants: From Screening up to Day 113
Arm/Group | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy | Normal Healthy Volunteer Cohort: Pooled Placebo | Cystic Fibrosis Cohort: ARO-ENaC 40 mg, Days 1-3, 22-24 | Cystic Fibrosis Cohort: Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/8 | 0/12 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 1/8 | 0/12 | 1/4 | 2/3
Other Adverse Events (participants affected / at risk) | 3/4 | 2/4 | 3/4 | 3/4 | 6/8 | 10/12 | 3/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 (N=4) | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 (N=4) | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 (N=4) | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 (N=4) | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy (N=8) | Normal Healthy Volunteer Cohort: Pooled Placebo (N=12) | Cystic Fibrosis Cohort: ARO-ENaC 40 mg, Days 1-3, 22-24 (N=4) | Cystic Fibrosis Cohort: Placebo (N=3)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Healthy Volunteer Cohort: ARO-ENaC 20 mg, Days 1-3 (N=4) | Normal Healthy Volunteer Cohort: ARO-ENaC 40 mg, Days 1-3 (N=4) | Normal Healthy Volunteer Cohort: ARO-ENaC 65 mg, Days 1-3 (N=4) | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 (N=4) | Normal Healthy Volunteer Cohort: ARO-ENaC 180 mg, Days 1-3 With Bronchoscopy (N=8) | Normal Healthy Volunteer Cohort: Pooled Placebo (N=12) | Cystic Fibrosis Cohort: ARO-ENaC 40 mg, Days 1-3, 22-24 (N=4) | Cystic Fibrosis Cohort: Placebo (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Application site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vascular access site bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vascular access site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 6 | 0 | 1
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
On 01 July 2021 a voluntary suspension of dosing by the Sponsor was initiated. All subjects who had completed all planned doses continued safety follow-up according to the scheduled activities. This suspension of dosing was due to preliminary findings in the 6-month chronic rat good laboratory practice (GLP) toxicology study. The voluntary suspension was unrelated to any safety findings in the AROENaC1001 study. Subsequent to this, the Sponsor decided to terminate the AROENaC1001 study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor retains first right to publish results for this multi-center study, and thereafter can review results communications prior to release and can embargo communications regarding trial results for a period that is 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication of results but can require removal of its confidential information (excluding results).

DOCUMENTS (2):
  • Study Protocol (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT04375514/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT04375514/SAP_001.pdf